CLINICAL TRIAL: NCT01330017
Title: A Randomized, Dose-ranging, Placebo-controlled Trial to Evaluate the Effects of Phenylephrine HCl Immediate Release Tablets on Nasal Congestion in Subjects With Seasonal Allergic Rhinitis
Brief Title: Effects of Phenylephrine on Nasal Congestion in Participants With Seasonal Allergic Rhinitis (P08156 AM2)(Completed)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18123; CL2010-06; P08156 (Other: Merck)
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Rhinitis; Seasonal Rhinitis
Keywords: Seasonal allergies
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic, Seasonal | interventions — Oxymetazoline; Loratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- PE 10 mg (Experimental)
  Interventions: Drug: Phenylephrine HCl; Drug: Placebo; Drug: Loratadine
- PE 20 mg (Experimental)
  Interventions: Drug: Phenylephrine HCl; Drug: Placebo; Drug: Loratadine
- PE 30 mg (Experimental)
  Interventions: Drug: Phenylephrine HCl; Drug: Placebo; Drug: Loratadine
- PE 40 mg (Experimental)
  Interventions: Drug: Phenylephrine HCl; Drug: Placebo; Drug: Loratadine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Loratadine

INTERVENTIONS:
Drug: Phenylephrine HCl — 10-mg immediate-release tablets, orally, up to 4 tablets per dose every 4 hours, for 7 days
  Other Names: SCH 002063
  Arms: PE 10 mg; PE 20 mg; PE 30 mg; PE 40 mg
Drug: Placebo — Placebo tablets, orally, up to five tablets per dose every 4 hours, for 7 days
Drug: Loratadine — 10-mg tablets, orally, once per day at a dose not to exceed 10 mg in a 24-hour period.
  Other Names: Claritin®

SUMMARY:
The trial will evaluate the nasal congestion symptom relief of the approved 10 mg phenylephrine (PE) dose and the higher 20 mg, 30 mg, and 40 mg PE doses compared with placebo in participants with histories of seasonal allergic rhinitis, using loratadine as background medication.

ELIGIBILITY:
Inclusion criteria:

* Female participants of reproductive potential must have a negative pregnancy test and agree to use acceptable methods of birth control throughout the study.
* Participant is willing to stop use of current decongestant and allergy medications during the trial.
* Participant has a documented or self-reported history of seasonal allergy.
* Participant has documented positive skin testing to spring pollen allergens.
* Participant has nasal congestion of at least moderate severity.
* Participant has mean seated (after 5 minutes of rest) systolic/diastolic blood pressure ≤138/88 mmHg.
* Participant has clinically acceptable physical exam and 12-lead electrocardiogram (ECG).
* Participant is without clinically significant disease.
* Participant must agree not to take monoamine oxidase inhibitor (MAOI) from 14 days before trial participation until 14 days after the end of the trial.
* Participant must sign an informed consent form

Exclusion criteria:

* Participants must not have any significant medical condition that is a contraindication to the use of phenylephrine HCl or loratadine, such as thyroid disease, uncontrolled diabetes mellitus, coronary heart disease, ischemic heart disease, elevated intraocular pressure, or prostatic hypertrophy.
* Participants with a history or presence of hypertension.
* Participants who have started allergen immunotherapy within a month preceding enrollment or starting allergen immunotherapy or anticipating immunotherapy dose change during the trial. Xolair (omalizumab) may not be used within 4 years prior to trial participation.
* Participants who have a known allergy or intolerance to phenylephrine HCl, any other decongestant, loratadine, desloratadine, or any other antihistamine.
* Participants with persistent asthma, rhinitis medicamentosa, or acute or chronic sinusitis, or a history of significant sinusitis within one month of enrollment.
* Participant with a history of intermittent asthma may be considered for enrollment provided they have no asthma symptoms at the time of enrollment and use only a short acting beta2-agonist less than twice weekly.
* Participants who have used systemic (oral, rectal, injectable), topical, or nasal corticosteroids in the last 30 days (up to 1% topical hydrocortisone is permitted).
* Participants using a leukotriene receptor antagonist for maintenance treatment of asthma.
* Participant with a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* Participant with a history of immunological disease or malignancy within the past 5 years, with the exception of non-melanoma skin cancer.
* Participant with positive drug screen (participants on prescribed medication resulting in a positive drug screen result may still be enrolled at the discretion of the investigator).
* Participant has had major surgery or participated in another investigational study within 4 weeks prior to the Screening Visit.
* Participants taking any herbal supplements during trial conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

REFERENCES:
- [Derived] Meltzer EO, Ratner PH, McGraw T. Oral Phenylephrine HCl for Nasal Congestion in Seasonal Allergic Rhinitis: A Randomized, Open-label, Placebo-controlled Study. J Allergy Clin Immunol Pract. 2015 Sep-Oct;3(5):702-8. doi: 10.1016/j.jaip.2015.05.007. Epub 2015 Jul 2. PMID 26143019

RESULTS

PARTICIPANT FLOW:
Groups:
- PE 10 mg: PE 10 mg was administered orally every 4 hours in combination with background loratadine treatment.
- PE 20 mg: PE 20 mg was administered orally every 4 hours in combination with background loratadine treatment.
- PE 30 mg: PE 30 mg was administered orally every 4 hours in combination with background loratadine treatment.
- PE 40 mg: PE 40 mg was administered orally every 4 hours in combination with background loratadine treatment.
- Placebo: Matching placebo was administered orally every 4 hours in combination with background loratadine treatment.
Period: Overall Study
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo
Started | 109 | 108 | 107 | 112 | 103
Completed | 104 | 104 | 99 | 100 | 100
Not Completed | 5 | 4 | 8 | 12 | 3
Not completed — Adverse Event | 0 | 1 | 1 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Unknown Reason | 5 | 3 | 5 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo | Total
Number analyzed (Participants) | 109 | 108 | 107 | 112 | 103 | 539
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (11.25) | 36.8 (11.08) | 38.9 (12.65) | 39.6 (13.10) | 38.9 (11.96) | 38.7 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 63 | 73 | 52 | 61 | 325
  Male | 33 | 45 | 34 | 60 | 42 | 214

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the Daily Reflective Nasal Congestion Score
Description: The reflective nasal congestion score was captured in participant diaries just before the 8:00 a.m. dose and 12 hours later just before the 8:00 p.m. dose. Participants rated congestion on a 4-point scale of severity from 0 (best) to 3 (worst), with 0 = absent symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms. The daily reflective nasal congestion symptom score was defined as the average of the morning and evening reflective nasal congestion score for the entire treatment period. Baseline was defined as the average of the daily scores over the 4 consecutive 24-hour periods before randomization.
Time Frame: Baseline, Day 7
Population: The Intent-to-Treat (ITT) population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Placebo: Matching placebo tablets were administered orally every 4 hours in combination with background loratadine treatment.
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo
Number analyzed (Participants) | 104 | 106 | 102 | 104 | 101
Units on a Scale | -0.460 (0.5374) | -0.499 (0.5042) | -0.508 (0.5618) | -0.461 (0.5308) | -0.428 (0.5530)
Statistical Analysis 1: Comparison: PE 10 mg vs Placebo; Test type: Superiority or Other; p = 0.4912, ANCOVA — The p-value reflects mean change from baseline vs. placebo from an ANCOVA model with adjustments for baseline reflective score value, investigative site, age, and gender
Statistical Analysis 2: Comparison: PE 20 mg vs Placebo; Test type: Superiority or Other; p = 0.4519, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: PE 30 mg vs Placebo; Test type: Superiority or Other; p = 0.2186, ANCOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: PE 40 mg vs Placebo; Test type: Superiority or Other; p = 0.5983, ANCOVA — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change From Baseline in the Morning (a.m.) Symptom Score for the Nasal Reflective Symptom Assessment by Study Day of the Treatment Period
Description: The morning reflective nasal congestion score was captured in participant diaries just before the 8:00 am dose. It is a composite score including four nasal symptoms: rhinorrhea, nasal congestion, nasal itching, and sneezing and it is rated on a 0-3 scale of severity with 0 = absent symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms.
Time Frame: Baseline and Days 2, 3, 4, 5, 6, and 7
Population: The ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo
Number analyzed (Participants) | 109 | 108 | 107 | 112 | 103
Units on a Scale
  Baseline (n = 109, 108, 106, 111, 102) | 2.417 (0.4327) | 2.517 (0.3995) | 2.481 (0.4148) | 2.492 (0.3887) | 2.514 (0.4208)
  Day 2 (n = 104, 106, 102, 104, 101) | -0.243 (0.6034) | -0.200 (0.5940) | -0.216 (0.6416) | -0.308 (0.6630) | -0.283 (0.6439)
  Day 3 (n = 104, 104, 102, 103, 101) | -0.359 (0.7750) | -0.362 (0.6883) | -0.324 (0.7109) | -0.369 (0.6679) | -0.362 (0.6834)
  Day 4 (n = 104, 104, 101, 102, 101) | -0.503 (0.7604) | -0.439 (0.7179) | -0.485 (0.7318) | -0.510 (0.7924) | -0.422 (0.7402)
  Day 5 (n = 104, 104, 101, 100, 100) | -0.426 (0.7881) | -0.458 (0.7118) | -0.465 (0.7365) | -0.474 (0.7762) | -0.392 (0.7236)
  Day 6 (n = 104, 104, 100, 100, 100) | -0.474 (0.7751) | -0.612 (0.8283) | -0.584 (0.7866) | -0.474 (0.7525) | -0.428 (0.7331)
  Day 7 (n = 104, 103, 100, 99, 100) | -0.541 (0.8543) | -0.472 (0.8186) | -0.594 (0.8256) | -0.539 (0.7858) | -0.438 (0.8296)

3. Secondary Outcome: Mean Change From Baseline in the Evening (p.m.) Symptom Score for the Nasal Reflective Symptom Assessment by Study Day of the Treatment Period
Description: The evening reflective nasal congestion score was captured in participant diaries just before the 8;00 p.m. dose. It is a composite score including four nasal symptoms: rhinorrhea, nasal congestion, nasal itching, and sneezing and is rated on a 0-3 scale of severity with 0 = absent, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms.
Time Frame: Baseline and Days 1, 2, 3, 4, 5, 6, and 7
Population: The ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo
Number analyzed (Participants) | 109 | 108 | 107 | 112 | 103
Units on a Scale
  Baseline (n = 109, 108, 106, 111, 102) | 2.376 (0.4521) | 2.361 (0.4577) | 2.363 (0.4514) | 2.362 (0.4476) | 2.380 (0.4846)
  Day 1 (n = 102, 106, 101, 102, 101) | -0.321 (0.6107) | -0.285 (0.5961) | -0.359 (0.7701) | -0.321 (0.6852) | -0.287 (0.7003)
  Day 2 (n = 102, 103, 102, 103, 101) | -0.360 (0.7240) | -0.410 (0.6650) | -0.483 (0.8177) | -0.466 (0.7646) | -0.386 (0.7988)
  Day 3 (n = 104, 104, 101, 101, 101) | -0.546 (0.7289) | -0.512 (0.7049) | -0.527 (0.8440) | -0.480 (0.7346) | -0.505 (0.7818)
  Day 4 (n = 104, 104, 101, 99, 100) | -0.536 (0.7524) | -0.474 (0.7479) | -0.597 (0.8653) | -0.533 (0.8227) | -0.450 (0.8142)
  Day 5 (n = 104, 102, 97, 99, 99) | -0.526 (0.7398) | -0.610 (0.7863) | -0.564 (0.9052) | -0.475 (0.7739) | -0.485 (0.8870)
  Day 6 (n = 104, 103, 100, 100, 100) | -0.613 (0.8539) | -0.750 (0.8105) | -0.648 (0.8624) | -0.597 (0.8704) | -0.470 (0.8515)
  Day 7 (n = 104, 102, 100, 98, 100) | -0.613 (0.7920) | -0.650 (0.7766) | -0.588 (0.9323) | -0.564 (0.7752) | -0.520 (0.8781)

4. Secondary Outcome: Mean Change From Baseline in the a.m. Symptom Score for the Instantaneous Nasal Symptom Assessment by Study Day of the Treatment Period
Description: Instantaneous assessment of nasal symptoms was performed once daily before the
  morning dose. The instantaneous assessment was a composite score of four nasal symptoms: rhinorrhea, nasal congestion, nasal itching, and sneezing and is rated on a 0-3 scale of severity with 0 = absent symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms.
Time Frame: Baseline and Day 2, 3, 4, 5, 6, and 7
Population: The ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo
Number analyzed (Participants) | 109 | 108 | 107 | 112 | 102
Units on a Scale
  Baseline (n = 107, 106, 104, 106, 101) | 2.271 (0.6669) | 2.311 (0.6527) | 2.298 (0.6809) | 2.311 (0.6228) | 2.406 (0.6030)
  Day 2 (n = 104, 105, 102, 103, 101) | -0.147 (0.6807) | 0.010 (0.7568) | -0.060 (0.7361) | -0.010 (0.6308) | -0.180 (0.7572)
  Day 3 (n = 104, 103, 102, 102, 101) | -0.265 (0.9002) | -0.206 (0.7491) | -0.130 (0.8246) | -0.112 (0.8234) | -0.130 (0.7740)
  Day 4 (n = 104, 103,101,101, 101) | -0.324 (0.8462) | -0.255 (0.8288) | -0.253 (0.9186) | -0.351 (0.8421) | -0.280 (0.8297)
  Day 5 (n = 104, 103, 101, 99, 101) | -0.304 (0.7550) | -0.314 (0.8672) | -0.283 (0.8456) | -0.232 (0.8927) | -0.240 (0.6980)
  Day 6 (n = 104, 104, 100, 99, 100) | -0.353 (0.8402) | -0.422 (0.9589) | -0.337 (0.8961) | -0.379 (0.8013) | -0.260 (0.7333)
  Day 7 (n = 104, 102, 100, 98, 100) | -0.382 (0.8330) | -0.376 (0.9258) | -0.408 (0.9176) | -0.404 (0.8591) | -0.380 (0.7625)

5. Secondary Outcome: Mean Change From Baseline for the Daily Reflective Nasal Symptom Assessment Score by Study Day of the Treatment Period
Description: The reflective nasal congestion score was captured in participant diaries just before the 8:00 a.m. dose and 12 hours later just before the 8:00 p.m. dose. It is a composite score including four nasal symptoms: rhinorrhea, nasal congestion, nasal itching, and sneezing and is rated on a 0-3 scale of severity with 0 = absent symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms. The daily reflective nasal congestion symptom score was defined as the average of the morning and evening reflective nasal congestion score for the entire treatment period.
Time Frame: Baseline and Days 1, 2, 3, 4, 5, 6, and 7
Population: The ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo
Number analyzed (Participants) | 109 | 108 | 107 | 112 | 103
Units on a Scale
  Baseline (n = 109. 108, 106, 111, 102) | 2.394 (0.3869) | 2.452 (0.3593) | 2.440 (0.3684) | 2.437 (0.3722) | 2.457 (0.4014)
  Day 1 (n = 102, 106, 101, 102, 101) | -0.353 (0.5821) | -0.367 (0.6130) | -0.431 (0.7168) | -0.389 (0.6408) | -0.364 (0.6125)
  Day 2 (n = 104, 106, 102, 104, 101) | -0.297 (0.5786) | -0.320 (0.5181) | -0.367 (0.5734) | -0.392 (0.5406) | -0.345 (0.6239)
  Day 3 (n = 104, 104, 102, 103, 101) | -0.451 (0.6566) | -0.449 (0.5989) | -0.441 (0.6548) | -0.425 (0.5806) | -0.444 (0.6383)
  Day 4 (n = 104, 104, 101, 102, 101) | -0.519 (0.6455) | -0.468 (0.6256) | -0.559 (0.6994) | -0.520 (0.7017) | -0.449 (0.6852)
  Day 5 (n = 104, 104, 101, 100, 101) | -0.475 (0.6831) | -0.550 (0.6478) | -0.529 (0.7278) | -0.484 (0.6992) | -0.444 (0.6859)
  Day 6 (n = 104, 104, 100, 100, 100) | -0.543 (0.7267) | -0.689 (0.7241) | -0.635 (0.6890) | -0.544 (0.7232) | -0.460 (0.6943)
  Day 7 (n = 104, 103, 100, 99, 100) | -0.576 (0.7385) | -0.573 (0.6821) | -0.610 (0.7658) | -0.556 (0.6695) | -0.490 (0.7770)

6. Secondary Outcome: Mean Change From Baseline for the Instantaneous Nasal Symptom Assessment Score By Study Day of the Treatment Period
Description: as for outcome 4
Time Frame: Baseline and Days 1, 2, 3, 4, 5, 6, and 7
Population: The ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo
Number analyzed (Participants) | 109 | 108 | 107 | 112 | 102
Units on a Scale
  Baseline (n = 107, 106, 104, 106, 101) | 2.271 (0.6669) | 2.311 (0.6527) | 2.298 (0.6809) | 2.311 (0.6228) | 2.406 (0.6030)
  Day 2 (n = 102, 104, 100, 99, 100) | -0.147 (0.6807) | 0.010 (0.7568) | -0.060 (0.7361) | -0.010 (0.6308) | -0.180 (0.7572)
  Day 3 (n = 102, 102, 100, 98, 100) | -0.265 (0.9002) | -0.206 (0.7491) | -0.130 (0.8246) | -0.112 (0.8234) | -0.130 (0.7740)
  Day 4 (n = 102, 102, 99, 97, 100) | -0.324 (0.8462) | -0.255 (0.8288) | -0.253 (0.9186) | -0.351 (0.8421) | -0.280 (0.8297)
  Day 5 (n = 102, 102, 99, 95, 100) | -0.304 (0.7550) | -0.314 (0.8672) | -0.283 (0.8456) | -0.232 (0.8927) | -0.240 (0.6980)
  Day 6 (n =102, 102, 98, 95, 100) | -0.353 (0.8402) | -0.422 (0.9589) | -0.337 (0.8961) | -0.379 (0.8013) | -0.260 (0.7333)
  Day 7 (n = 102, 101, 98, 94, 100) | -0.382 (0.8330) | -0.376 (0.9258) | -0.408 (0.9176) | -0.404 (0.8591) | -0.380 (0.7625)

7. Secondary Outcome: Time to Maximal Effect
Description: Time to maximal effect is defined as the earliest time that the nasal congestion symptom score demonstrates the greatest numerical difference from the placebo in change from baseline. The mean change from baseline scores for a treatment arm and for the placebo arm at each day and timepoint of the treatment period (Day 1 morn, Day 1 eve, etc) were calculated. Then the difference between the placebo and treatment arm means at each day/timepoint of the treatment period was calculated and recorded the day/timepoint that the difference between the treatment arm and the placebo was highest.
Time Frame: Baseline up to Day 7
Population: The ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Days
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg
Number analyzed (Participants) | 109 | 108 | 107 | 112
Days | 5.5 | 5.5 | 5.5 | 5.5

8. Secondary Outcome: Change From Baseline for the Instantaneous Nasal Symptom Assessment Score at Day 7
Description: The magnitude of effect was measured as the change from baseline for the instantaneous nasal symptom assessment score at Day 7. Instantaneous assessment of nasal symptoms was performed once daily before the morning dose. The instantaneous assessment was a composite score of four nasal symptoms: rhinorrhea, nasal congestion, nasal itching, and sneezing and is rated on a 0-3 scale of severity with 0 = absent symptoms, 1 = mild symptoms, 2 = moderate symptoms, and 3 = severe symptoms.
Time Frame: Baseline, Day 7
Population: The ITT population included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo
Number analyzed (Participants) | 102 | 101 | 98 | 94 | 100
Units on a Scale | -0.382 (0.8330) | -0.376 (0.9258) | -0.408 (0.9176) | -0.404 (0.8591) | -0.380 (0.7625)

ADVERSE EVENTS:
Arm/Group | PE 10 mg | PE 20 mg | PE 30 mg | PE 40 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/108 | 0/107 | 1/112 | 0/103
Other Adverse Events (participants affected / at risk) | 6/109 | 4/108 | 3/107 | 3/112 | 0/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PE 10 mg (N=109) | PE 20 mg (N=108) | PE 30 mg (N=107) | PE 40 mg (N=112) | Placebo (N=103)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PE 10 mg (N=109) | PE 20 mg (N=108) | PE 30 mg (N=107) | PE 40 mg (N=112) | Placebo (N=103)
Headache (Nervous system disorders) | 6 (6) | 4 (4) | 3 (3) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission or publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.